CLINICAL TRIAL: NCT01794039
Title: Randomized Phase 2 Trial of Retreatment With Pomalidomide or Lenalidomide With Dexamethasone for Patients With Relapsed Myeloma
Brief Title: Pomalidomide or Lenalidomide and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma Previously Treated With Lenalidomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1187; NCI-2013-00412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-006426; MCCC Add 1; MC1187 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (lenalidomide, dexamethasone) (Experimental): Patients receive lenalidomide PO daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may crossover to arm B.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide
- Arm B (pomalidomide, dexamethasone) (Experimental): Patients receive pomalidomide PO daily on days 1-21 and dexamethasone as in arm A. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm A (lenalidomide, dexamethasone)
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Pomalyst
  Arms: Arm B (pomalidomide, dexamethasone)

SUMMARY:
This randomized phase II trial studies how well pomalidomide and dexamethasone work compared to lenalidomide and dexamethasone in treating patients with multiple myeloma that has returned after a period of improvement (relapsed) or did not respond to previous treatment with lenalidomide (refractory). Pomalidomide and lenalidomide may help the immune system kill cancer cells and may also prevent the growth of new blood vessels that tumors need to grow. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dexamethasone may also help pomalidomide and lenalidomide work better by making cancer cells more sensitive to the drugs. It is not yet known whether pomalidomide and dexamethasone or lenalidomide and dexamethasone are effective in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the confirmed response rate of the combination of lenalidomide and dexamethasone in patients with relapsed myeloma who have previously become refractory to lenalidomide. (Arm A) II. To assess the confirmed response rate of the combination of pomalidomide and dexamethasone in patients with relapsed myeloma who have previously become refractory to lenalidomide. (Arm B)

SECONDARY OBJECTIVES:

I. To assess the toxicity in each arm in patients with relapsed myeloma who have previously received lenalidomide.

II. To assess the response rates with pomalidomide and dexamethasone in patients relapsing on lenalidomide and dexamethasone. (Arm A) III. To assess time to progression and overall survival with each approach.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive lenalidomide orally (PO) daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may crossover to arm B.

ARM B: Patients receive pomalidomide PO daily on days 1-21 and dexamethasone as in arm A. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Calculated creatinine clearance >= 30 ml/min by Cockcroft-Gault formula
* Absolute neutrophil count >= 1000uL
* (Untransfused) platelet count >= 50000/uL
* Hemoglobin >= 8.0 g/dL
* Relapsed myeloma that previously became refractory to lenalidomide, after initial response of partial response or better to the drug; refractory is defined as progression on treatment with a dose of at least 10 mg daily for lenalidomide; greater than or equal to 180 days must have elapsed since previous lenalidomide therapy was stopped
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Previously treated; NOTE: no limit to prior therapy provided there is adequate residual organ function
* Provide informed written consent
* Females of childbearing potential (FCBP)* must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days as required by Revlimid Risk Evaluation and Mitigation Strategy [REMS]), and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all study participants must be registered into the Revlimid REMS program, and be willing and able to comply with the requirements of Revlimid REMS program

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Willing to return to Mayo Clinic enrolling institution for follow-up

Exclusion Criteria:

* Residual toxicity of > grade 1 from prior therapy
* Other active malignancy < 1 year prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Any of the following:

  * Pregnant women
  * Nursing women (lactating females must agree not to breast feed while taking lenalidomide)
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* New York Heart Association classification III or IV
* Diagnosed active deep vein thrombosis (DVT) that has not been therapeutically anticoagulated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Lenalidomide, Dexamethasone): Patients receive lenalidomide PO daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may crossover to arm B.> > Dexamethasone: Given PO>
  > Lenalidomide: Given PO
- Arm B (Pomalidomide, Dexamethasone): Patients receive pomalidomide PO daily on days 1-21 and dexamethasone as in arm A. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.> > Dexamethasone: Given PO>
  > Pomalidomide: Given PO
Period: Overall Study
Arm/Group | Arm A (Lenalidomide, Dexamethasone) | Arm B (Pomalidomide, Dexamethasone)
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Lenalidomide, Dexamethasone) | Arm B (Pomalidomide, Dexamethasone) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Median (Full Range); unit: years] | 67 [64 to 75] | 68.5 [60 to 72] | 67 [60 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Tumor Responses Defined to be a Partial Response or Better Noted as the Objective Status on Two Consecutive Evaluations
Description: The proportion of successes will be estimated in each arm independently by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. A confirmed tumor response is defined to be a partial response or better noted as the objective status on two consecutive evaluations while receiving lenalidomide and dexmethasone (Arm A) or pomalidomide and dexamethasone (Arm B). All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.The International Myeloma Working Group (IMWG) uniform response criteria (Rajkumar et al, 2011) will be used to assess response to therapy.
Time Frame: Up to 2 years
Population: All patients that received treatment were evaluable for response
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm A (Lenalidomide, Dexamethasone): Patients receive lenalidomide PO daily on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing progressive disease may crossover to arm B.
  >
  > Dexamethasone: Given PO
  >
  > Lenalidomide: Given PO
- Arm B (Pomalidomide, Dexamethasone): Patients receive pomalidomide PO daily on days 1-21 and dexamethasone as in arm A. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Dexamethasone: Given PO
  >
  > Pomalidomide: Given PO
Arm/Group | Arm A (Lenalidomide, Dexamethasone) | Arm B (Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 5 | 4
proportion of participants | .4 [.05 to .85] | .25 [.006 to .81]

2. Secondary Outcome: Number of Participants With Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns. These results are reported in the Adverse Events section of this CT.gov report.
Time Frame: Up to 30 days after last day of study drug treatment
Population: All treated patients are evaluable for Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Lenalidomide, Dexamethasone) | Arm B (Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 5 | 4
Participants | 5 | 4

3. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier. Due to an early closer from slow accrual the data from both arms was combined in survival analysis.
Time Frame: Time from registration to death due to any cause, assessed up to 2 years
Population: All patients that received Arm A or Arm B treatment.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arms A and B: 4 arm A patients were transferred to Arm B for further treatment. Arm A patients, that went off study for any reason, were allowed to transfer to Arm B.
Arm/Group | Arms A and B
Number analyzed (Participants) | 9
Months | 13.4 [9.3 to NA] — Upper confidence interval was not reached

4. Secondary Outcome: Time to Progression
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier. The International Myeloma Working Group (IMWG) uniform response criteria (Rajkumar et al, 2011) will be used to assess response to therapy.
Time Frame: Time from registration to the earliest date with documentation of disease progression, assessed up to 2 years
Population: All patients that received Arm A or Arm B treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arms A and B
Number analyzed (Participants) | 9
Months | 10 [4.1 to 12.4]

ADVERSE EVENTS:
Arm/Group | Arm A (Lenalidomide, Dexamethasone) | Arm B (Pomalidomide, Dexamethasone)
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Lenalidomide, Dexamethasone) (N=5) | Arm B (Pomalidomide, Dexamethasone) (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Lenalidomide, Dexamethasone) (N=5) | Arm B (Pomalidomide, Dexamethasone) (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 1 (2)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (5) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 4 (23) | 2 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (4) | 2 (5)
Fatigue (General disorders) | 5 (36) | 3 (15)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (25) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (18) | 2 (7)
Platelet count decreased (Investigations) | 4 (30) | 2 (7)
White blood cell decreased (Investigations) | 5 (24) | 3 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (46) | 3 (15)
Tremor (Nervous system disorders) | 0 (0) | 1 (9)
Agitation (Psychiatric disorders) | 1 (5) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes